CLINICAL TRIAL: NCT02187237
Title: A RandomizEd DoUble Blinded Controlled Study to Evaluate the Safety and Effectiveness of the "YOLO TOUCH" Low Level Laser Therapy (LLLT) for Circumference Reduction of he Waistline - REDUCE
Brief Title: Safety and Effectiveness of the "YOLO TOUCH" LLLT for Circumference Reduction of the Waistline
Acronym: REDUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yolo Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: YTCSP-2013-YOLO-REDUCE
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Reduction of the Waist Circumference

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser therapy (Experimental)
  Interventions: Device: YOLO TOUCH Low Level Laser

INTERVENTIONS:
Device: YOLO TOUCH Low Level Laser

SUMMARY:
The YOLO TOUCH consists of a console and multi-probes that are placed on the treatment area that emit laser light to reduce the circumference waistline.

DETAILED DESCRIPTION:
The YOLO TOUCH device is class II device intended for use in circumference reduction of the waist as a non-invasive, non-thermal, and low energy laser. Typical area of the body for use with the YOLO TOUCH is the abdominal area.

The YOLO TOUCH low-level therapy device consists of a main console and 8 multi-probes that are constructed so that each probe contains 12 laser emission diode sources at a power output of 35mW per diode.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult ≥ 18 years old and <65 years of age
* Subject has maintained a stable weight for the past 6 months (variation no greater than 10 lbs. from "usual weight")
* Subject is willing to maintain current diet and exercise regimen for the duration of the study.
* Subject is willing and able to provide written informed consent.
* Subject is willing to return for all scheduled and required visits.
* Subject is willing to comply with post-laser treatment cardiovascular exercise.
* Subject is willing to comply with food and fluid requirements pre-treatment and post-treatment.

Exclusion Criteria:

* Subject is on an active weight control regimen.
* Subject has a pacemaker.
* Subject has a history of epilepsy.
* Subject has a history of any type of cancer, including skin cancer.
* Subject had a prior surgical intervention for body sculpting/weight loss such as liposuction, abdominoplasty, gastroplasty, lap band surgery, etc.
* Subject has a medical, physical, or other contraindications for body sculpting/weight loss.
* Subject has an active infection, wound or other external trauma to the areas to be treated with the laser.
* Subject is pregnant, breast feeding, or planning pregnancy prior to study end.
* Subject is participating in any treatment other than the study procedure (existing or new) to promote body contouring and/or weight loss during the course o the study participation.
* Subject is participating in another research study of a device, medication, biologic, or other agent within 30 days or could, in the opinion of the investigator, affect the results of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Reduction of girth measurements for the waistline | 3 weeks
  Reduction of one (1.0) inch of girth measurement in the average of three circumference measurements for the waistline from baseline to after completion of the three (3) week study procedure (i.e., after nine (9) twenty (20) minute laser treatments - three (3) per week for three (3) weeks.

SECONDARY OUTCOMES:
Complications, device related adverse events during LLLT and device related adverse events post LLLT. | up to at day 50

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Portz, M.D., Principal Investigator — Burnett Sports Perfomance Center
Locations (1):
- Burnett Sports Performance Center, McMurray, Pennsylvania, United States